CLINICAL TRIAL: NCT03223116
Title: Radiofrequency Energy Delivery for Gastroesophageal Reflux Disease: A Prospective, Multicenter Clinical Trial From China
Brief Title: Radiofrequency Energy Delivery for Gastroesophageal Reflux Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director, Head of Department of Gastroenterology, Principal Investigator, Clinical Professor, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC2015
Record Dates: First submitted 2017-06-30; First posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: heartburn; regurgitation
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiofrequency (Experimental): Radiofrequency delivery to the gastroesophageal junction
  Interventions: Procedure: Radiofrequency delivery

INTERVENTIONS:
Procedure: Radiofrequency delivery — Radiofrequency to the gastroesophageal junction

SUMMARY:
This study is to evaluate the safety and efficacy of radiofrequency energy procedure for Gastro-esophageal reflux disease (GERD) based on changes of symptoms, medication esophagitis grade, esophageal acid exposure and lower esophageal sphincter pressure. Symptom assessment was performed at baseline and 3, 6, 12 months after treatment.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is a chronic disease characterized by symptoms of heartburn and acid regurgitation. Uncontrolled GERD can significantly impact quality of life. The use of proton pump inhibitors (PPI) remains the mainstay therapy. However, the efficacy of this intervention is often hampered by adherence, costs, and the risks of long-term PPI use. Anti-reflux surgery is an option for patients with refractory symptoms or in those in whom medical therapy is contraindicated or not desirable, but the incidence of dysphagia, abdominal distension associated wth the surgery is high. Radiofrequency ablation, minimally invasive, less complications, has become alternative treatments options. But the current research on radiofrequency treatment of the data is limited in China. Therefore, the investigators conduct this multi-center clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* diagnosis of GERD established by either

  * 24-h oesophageal pH monitoring (performed off medications) showing an abnormal OAE (pH < 4 at least 4% of time) and/or
  * an upper gastrointestinal (GI) endoscopy showing oesophagitis grade A or B in Los Angeles (LA) classification
* presence of typical symptoms of GERD (heartburn and ⁄or regurgitation with at least three episodes of typical symptoms per week in the absence of PPI therapy),
* adequate symptom relief obtained with PPIs,but needing maintenance with at least standard dose.

Exclusion Criteria:

* presence of Barrett's oesophagus >3 cm and ⁄or with dysplasia and ⁄or previously treated,
* presence of hiatus hernia >3 cm,
* presence of oesophagitis grade C or D in LA classification,
* presence of oesophageal stricture or achalasia,
* history of oesophageal or gastric surgery,
* presence of gastric or oesophageal varices,
* impossibility to stop an anticoagulant therapy or severe coagulopathy,
* any contraindication to general anaesthesia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-09-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline GERD-HRQL scores at 12 months | 12 months
  Assess the GERD-HRQL scores at 12 month and compare it with the baseline

SECONDARY OUTCOMES:
Change from baseline esophagitis grade at 12 months | 12 months
  Assess the esophagitis condition at 12 month and compare it with the baseline
Change from baseline esophageal acid exposure times from at 12 months | 12 month
  Measure the esophageal acid exposure at 12 months and compare it with the baseline
Change from baseline lower esophageal sphincter pressure at 12 months | 12 month
  Measure the lower esophageal sphincter pressure at 12 month and compare it with the baseline
Change from baseline medication at 12 months | 12 months
  Assess dosage of the medication at 12 month and compare it with the baseline

CONTACTS AND LOCATIONS:
Overall Officials: zhaoshen Li, MD, Study Chair — Changhai Hospital
Locations (1):
- Departmentof Gastroenterology Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fock KM, Talley N, Goh KL, Sugano K, Katelaris P, Holtmann G, Pandolfino JE, Sharma P, Ang TL, Hongo M, Wu J, Chen M, Choi MG, Law NM, Sheu BS, Zhang J, Ho KY, Sollano J, Rani AA, Kositchaiwat C, Bhatia S. Asia-Pacific consensus on the management of gastro-oesophageal reflux disease: an update focusing on refractory reflux disease and Barrett's oesophagus. Gut. 2016 Sep;65(9):1402-15. doi: 10.1136/gutjnl-2016-311715. Epub 2016 Jun 3. PMID 27261337